CLINICAL TRIAL: NCT01723059
Title: Conventional Therapy vs Sequential Therapy for the Treatment of Helicobacter Pylori Infection
Brief Title: Standard Triple Therapy vs Sequential Therapy in Treatment of H Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Principal Investigator, Byron Cryer, Staff Gastroenterologist, Dallas VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-060
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Helicobacter Infection
MeSH Terms: conditions — Helicobacter Infections | interventions — Amoxicillin; Omeprazole; Clarithromycin; technetium Tc 99m 1,6-di-(2-thienyl)-2,5-diazahexane; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard triple therapy (Other): Gold standard for management of H pylori is amoxicillin 1 gm twice daily, clarithromycin 500 mg twice daily, and omeprazole 20 mg twice daily for 10 days.
  Interventions: Drug: Standard Triple Therapy
- Sequential Therapy (Active Comparator): Amoxicillin 1 gm twice daily and omeprazole 20 mg twice daily for 5 days followed by metronidazole 500 mg twice daily, clarithromycin 500 mg twice daily, and omeprazole 20 mg twice daily for 5 days.
  Interventions: Drug: Sequential Therapy

INTERVENTIONS:
Drug: Standard Triple Therapy — for 10 days
  Other Names: Amoxicillin 1000 mg orally twice daily; Omeprazole 20 mg orally twice daily; Clarithromycin 500 mg orally twice daily
  Arms: Standard triple therapy
Drug: Sequential Therapy — total 10 days
  Other Names: Amoxicillin 1000 mg orally twice daily for 5 days; Omeprazole 20 mg orally twice daily for 5 days; Then; Clarithromycin 500 mg orally twice daily for 5 days; Metronidazole 500 mg orally twice daily for 5 days
  Arms: Sequential Therapy

SUMMARY:
Traditionally, H pylori infection has been treated with conventional triple therapy. This includes amoxicillin, clarithromycin and a proton pump inhibitor all given daily for 10-14 days. In Europe, the guidelines now advocate treatment of H pylori with sequential therapy which is 5 days of amoxicillin therapy with proton pump inhibitor followed by 5 days of clarithromycin, metronidazole, and proton pump inhibitor with better response rates. We hypothesize that H. pylori resistance pattern and treatment response rates observed in Europe will not be predictive of resistance patterns and response rates in the United States.

ELIGIBILITY:
Inclusion Criteria:

Subject has signed informed consent Subject is an adult older than 18 yrs old and requires an upper endoscopic evaluation If female and of child bearing potential, subject has a negative pregnancy test and is not nursing.

Patient has not received prior treatment for H pylori Subject is able to understand and comply with study procedures

Exclusion Criteria:

Recent use (within 4 weeks) of any of the medications used in the treatment of H pylori(Amoxicillin, Clarithromycin, Metronidazole) Subject undergoing endoscopy for acute gastrointestinal bleeding Subject has an allergy to any of the medications used in the treatment of H pylori Subject has a history of esophageal or gastric carcinoma including lymphoma Subject has esophageal varices or undergoing endoscopy for esophageal banding Subject is taking warfarin or clopidogrel Subject has coagulopathy that precludes safe biopsy of the biopsy areas Subject has comorbidity that precludes safe participation in the study Subject is a pregnant female Subject has a history of H. pylori infection. Patient is already enrolled in GI Study. History of UGI surgery other than Nissen Fundoplication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 4 weeks after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Byron Cryer, MD, Principal Investigator — Gastroenterologist, MD VA; Robert Genta, MD, Study Chair — Pathologist, MD; Elizabeth Coss, MD, Study Chair — Gastroenterology Fellow, MD
Locations (1):
- Dallas VAMC, Dallas, Texas, United States